CLINICAL TRIAL: NCT06116773
Title: Effectiveness of Early Cardiac Rehabilitation After Coronary Artery Bypass Graft Surgery
Brief Title: Effectiveness of Early Cardiac Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Raziye Ceylan, master of science, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-RC-01
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: Early Cardiac Rehabilitation; Coronary Artery Bypass Graft Surgery; Functional Capacity; Quality of Life; Frailty
MeSH Terms: conditions — Coronary Artery Disease; Frailty

STUDY DESIGN:
Intervention Model Description: two groups: training group and control group.
Who Masked: Outcomes Assessor
Masking Description: our study was conducted as single (assessor) blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Training group, in addition to secondary prevention approaches and home exercise program, will be applied 3 sessions/week, 60 minutes of supervised cardiac rehabilitation program for 8 weeks.
  Interventions: Other: Training
- Control Group (Active Comparator): Control group will be informed about secondary prevention approaches and a home exercise program will be recommended.
  Interventions: Other: Control

INTERVENTIONS:
Other: Training — Training group is supervised exercise group and will be included in a supervised cardiac rehabilitation program for 3 days a week. The program will start 2 weeks after CABG surgery and continue for 8 weeks, totaling 24 sessions. Aerobic, resistance, balance and stretching exercises will be applied within the program. Total exercise time is aimed to be ≥150 min/week for 8 weeks. A home-based exercise program will be recommended.
  Moderate-intensity continuous aerobic training will be implemented using an upright exercise bike (5 minutes warm-up, 20 minutes load, 5 minutes cool down, 5 minutes recovery). Rhythmic unloaded aerobic exercises or low-load (0.5-1 kg) resistance exercises (starting from the 6th week post-op) will be performed for an average of 15-20 minutes. Balance exercises will progress from easy to difficult depending on the person's performance. Stretching exercise for the gastrocnemius muscle will be performed for 4 repetitions in a short stretching period of 15 seconds.
  Arms: Training Group
Other: Control — Patients will be informed about secondary prevention approaches which is routinely performed after discharge after CABG operation and will be recommended a home-based exercise program. Patients will be called by phone once a week and exercise monitoring will be provided. Recommended home exercise program includes:
  * Breathing exercises
  * Moderate intensity (RPE 4-6) walking (150 min/week).
  * Posture exercises (shoulder elevation-depression, 90 degree shoulder flex-extend, 90 degree shoulder abd-add, neck joint range of motion exercises)
  * They will be advised to continue range of motion exercises in the early post-operative period. (Twice a day, 10 repetitions).These exercises include ankle dorsi-plantar flexion, hip abduction-adduction, hip internal-external rotation, hip flexion-extension, arm elevation-depression in the supine position; flexion-extension in the sitting position; hip abduction-adduction, hip hyperextension and counting movements in the standing position.
  Arms: Control Group

SUMMARY:
The goal of this experimental study is to compare the effects of early (2nd week) cardiac rehabilitation applied in addition to usual care on functional capacity, quality of life, frailty and body composition in patients undergoing coronary artery bypass graft surgery.

The main questions it aims to answer are:

* Does early cardiac rehabilitation contribute to increasing functional capacity?
* Does early cardiac rehabilitation have positive effects on quality of life, frailty and body composition?

Participants will be divided into 2 groups (n = 50) in a randomized controlled manner. Patients in the training group (n:25) will participate in an 8-week supervised cardiac rehabilitation program as an outpatient after discharge. Patients in the control group (n:25) will be provided with usual care after discharge.

The control group will be informed about secondary prevention approaches and a home-based exercise program will be recommended. In addition to secondary prevention approaches and home-based exercise program, the training group will receive 3 sessions/week, 60 minutes of supervised cardiac rehabilitation for 8 weeks. All patients will be evaluated at baseline and after 8 weeks.

Researchers will compare training and control groups to see if effects on functional capacity, quality of life, frailty, body composition

DETAILED DESCRIPTION:
Cardiovascular diseases are still the number one cause of death worldwide, despite significant advances in diagnosis and treatment over the last 50 years. Coronary artery bypass graft (CABG) surgery is an important treatment option for coronary heart disease. Cardiac rehabilitation (CR) programs are a planned multidisciplinary approach to supervise exercise and educate patients about coronary artery disease risk factors and disease management. Cardiac rehabilitation consists of 3 main phases: in-hospital period (phase 1); early post-discharge period (phase 2) and exercise training period (phase 3). Cardiac rehabilitation phase II (KRII) is a secondary prevention program designed to restore health following a cardiac event and reduce the risk of mortality and future cardiac events. It covers approximately 2-12 weeks after discharge. This is the period when patients are closely monitored. A gradual physical activity program is applied according to the results of the applied tests. Participation in KRII is known to reduce hospital readmissions and mortality. Referral to KRII following an acute cardiac event is a Class IA recommendation.

Outpatient CR programs are designed to reduce the deconditioning negative effects of medical and surgical interventions in cardiac patients and have well-accepted health and survival benefits. CR improves exercise capacity, quality of life, and long-term prognosis in patients with coronary artery disease. The beneficial effects of cardiac rehabilitation applied to patients after CABG surgery on exercise capacity, coronary risk factors and quality of life have been documented (PubMed identification (ID): 22064600). Positive benefits of postdischarge exercise training have been demonstrated (PubMed ID: 10961975), and it seems reasonable to begin exercise training immediately after CABG surgery (PubMed ID: 23851406). A recent multicenter study showed that patients who actively participated in an outpatient CR program after CABG surgery exhibited greater improvement in exercise capacity and better survival without cardiovascular events than those who did not participate in the CR program (PubMed ID: 32037378).

Prior to this, international guidelines did not recommend resistance training as part of the CR program immediately after CABG surgery, with the rationale that physical exertion causes pressure or stress in the sternal area and should therefore be avoided for at least 6 weeks and 3 months after surgery. However, results of a published meta-analysis (PubMed ID: 20482475) suggest that resistance training is an effective exercise program to improve 6-minute walking distance in individuals with chronic heart failure.

The goals of resistance training in older adults are to increase exercise and functional capacity, reduce activity limitation, and improve functionality in performing daily activity, thereby improving social reintegration and health-related quality of life. Resistance training in older adults may increase muscle strength and endurance and thus prevent age-related loss of skeletal muscle mass and strength as well as loss of bone mass. Strength and balance are closely related and are important in improving dynamic balance and increasing strength, which helps maintain activities of daily living and prevent frailty in very old adults. Studies have been conducted to evaluate the effects of combined aerobic and resistance training on the functional capacity of patients undergoing CABG surgery. Studies (PubMed ID: 19477380, PubMed ID: 19782265) showed that combined training caused a significant improvement in peak oxygen uptake in this patient population. While CR is recommended to begin as soon as possible after discharge, enrollment typically occurs several weeks after hospital discharge. This creates a gap in rehabilitative care. Reduced physiological reserve resulting from surgery, hospitalization, and the recovery period between discharge and CR may increase the risk of postoperative complications, readmission, and physical disability. It is known that a delay in starting CR prolongs recovery, increases dependency on family/caregivers, and especially those of working age are negatively affected. Additionally, any delay may reduce the benefits of KR.

Many patients rapidly lose muscle and bone mass during sedentary periods after sternotomy, increasing the risk of falls and prolonging recovery time. Accordingly, a number of preliminary studies have shown superior results when activity is started earlier after sternotomy. (PubMed ID: 26722187, PubMed ID: 28101566, PubMed ID: 29602750, PubMed ID: 31504913). A current study also proved that starting exercise training 2 weeks after sternotomy is effective and safe (PubMed ID: 35731506 ).With this study plan, we hypothesized that comprehensive cardiac rehabilitation in the early period after CABG would increase functional capacity. The aim of our study is to investigate the effectiveness of early (2nd week) phase 2 cardiac rehabilitation compared to usual care in patients undergoing CABG surgery, based on the primary outcome of functional capacity and secondary outcomes of quality of life, frailty, and body composition. This study will be an important study investigating the effects of phase 2 cardiac rehabilitation applied in the early period (2nd week) after CABG surgery on functional capacity, quality of life, fragility and body composition.

ELIGIBILITY:
Inclusion Criteria:

* ⩾65 years old patients who underwent CABG surgery in the 2nd week post-op
* No contraindications for exercise training and ability to exercise
* Patients without diagnosed cognitive impairment

Exclusion Criteria:

* Cardiac arrhythmias that pose a serious risk
* Unstable angina
* Decompensated heart failure
* Unstable blood pressure control
* Peripheral artery disease with claudication
* Severe myocardial ischemia
* Cerebrovascular disease
* Orthopedic disease
* Chronic kidney disease (creatinine >3.0 mg/dL)
* Liver dysfunction (alanine aminotransferase >200 U/L)
* Other serious organ failure and/or other medical causes (e.g. difficulty walking)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Six minute walk test (6MWT) | eight weeks
  Functional capacity will be evaluated with the 6-minute walk test (6MWT). Patients will be walked in a 30-meter-long corridor for 6 minutes and the maximum walking distance will be measured. Before and after the test, heart rate, blood pressure and O2 saturation will be measured with pulse oximetry, and dyspnea and fatigue levels will be determined according to the Modified Borg scale.

SECONDARY OUTCOMES:
Modified Borg Scale | eight weeks
  Modified Borg Scale is used to determine the level of dyspnea and fatigue at rest and with exertion. Dyspnea and fatigue levels before and after 6 WT will be evaluated with the 'Modified Borg Dyspnea' and 'Modified Borg Fatigue' scales. These scales are subjective scales. In addition to being frequently used to determine the severity of dyspnea and fatigue observed with exertion, they are also suitable for the evaluation of dyspnea and fatigue at rest. They consist of ten items that indicate the severity of dyspnea and fatigue according to their degree. Scoring is made between 0: none at all - 10: very severe.
New York Heart Association (NYHA) functional classification | eight weeks
  Patients are classified from I to IV according to their physical activities. It is a strong prognosis indicator and risk marker. As the functional class increases, the survival rate decreases.
Modified Medical Research Council (MMRC) dyspnea scale | eight weeks
  It is used to assess dyspnea. MMRC is a scale developed to evaluate the dyspnea degree of patients more objectively. 5 points include activities that provoke a feeling of breathlessness, such as walking and climbing stairs. In less than a minute, the patient chooses a score from the MMRC scale based on his/her degree of dyspnea. The MMRC scale is defined as a differential tool that categorizes patients according to their disease levels.
Frail Scale | eight weeks
  It is used to assess frailty. It consists of 5 items; fatigue state, resistance, mobility, weight loss, and existing diseases. Depending on the answer given by the patients, a score of zero or one is given. Patients with a total score of zero are considered non-frail, 1-2 points are considered pre-frail, and patients with >2 points are considered frail.
Short Physical Performance Battery | eight weeks
  It consists of 3 objective tests that evaluate balance, walking speed and chair rising performance.
  Each test is scored between 0 (inability to complete the test) and 4 (highest level of performance). The scores from all three tests are summed to obtain a total score of 0-12. For a diagnosis of frailty, a total score of ≤5/12 is expected.
  4 Meter Walking Test: The person is asked to walk at normal walking speed for 4 meters.
  Five Times Sit to Stand Test: The person is asked to sit on the chair and stand up 5 times as quickly as possible and without stopping, crossing his arms on his chest, and the time elapsed when the fifth repetition is completed is recorded.
  Balance Tests: For static balance assessment, the person is asked to maintain 3 different standing postures (feet side by side, semi-tandem and tandem positions), which gradually become more difficult, for 10 seconds.
Mac New Heart Disease Health-Related Quality of Life Questionnaire | eight weeks
  It is a scale developed to determine the quality of life in heart diseases, consisting of 27 items, each with a 7-point Likert-type response. Three sub-groups (emotional, physical and social) and total score values are used in the evaluation of the scale.
  When calculating the scores for the sub-groups and the overall scale, the averages of the items in each dimension are taken. Therefore, scores range from 1 to 7 on average. A low score indicates worse quality of life, a high score indicates better quality of life.
Muscle strength | eight weeks
  The hand grip strength measurement test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer is used to perform the test.
  Grip strength should be assessed while the patient is sitting in a chair. Elbows are kept close to the body and 90° flexed. The wrist is in neutral. The person to be measured is asked to grasp the dynamometer and squeeze it as hard as he can. The test result is determined by calculating the average of three measurements.
Body composition | eight weeks
  It will be determined using a multifrequency bioelectric body impedance analysis (BIA) device. All measurements are taken in the morning and with as little clothing as possible. Participants are informed to urinate before measurement, not to engage in heavy physical activity within 12 hours, not to drink alcohol in the last 24 hours, and not to consume anything solid or liquid in the last 3 hours. After the participants' height and age information are entered into the software, they are asked to step on the aluminum insoles on the bottom of the device and hold the handles. As a result of the evaluation, the body Weight (kg), body mass index (BMI, kg/m2), fat percentage, muscle weight (kg), fluid percentage and amount of internal fat (kg) are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof, Study Director — Istanbul University - Cerrahpasa; Raziye Ceylan, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):2610-42. doi: 10.1161/CIR.0b013e31823b5fee. Epub 2011 Nov 7. No abstract available. PMID 22064600
- [Background] Balady GJ, Ades PA, Comoss P, Limacher M, Pina IL, Southard D, Williams MA, Bazzarre T. Core components of cardiac rehabilitation/secondary prevention programs: A statement for healthcare professionals from the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation Writing Group. Circulation. 2000 Aug 29;102(9):1069-73. doi: 10.1161/01.cir.102.9.1069. No abstract available. PMID 10961975
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Origuchi H, Itoh H, Momomura SI, Nohara R, Daida H, Masuda T, Kohzuki M, Makita S, Ueshima K, Nagayama M, Omiya K, Adachi H, Goto Y. Active Participation in Outpatient Cardiac Rehabilitation Is Associated With Better Prognosis After Coronary Artery Bypass Graft Surgery - J-REHAB CABG Study. Circ J. 2020 Feb 25;84(3):427-435. doi: 10.1253/circj.CJ-19-0650. Epub 2020 Feb 8. PMID 32037378
- [Background] Hwang CL, Chien CL, Wu YT. Resistance training increases 6-minute walk distance in people with chronic heart failure: a systematic review. J Physiother. 2010;56(2):87-96. doi: 10.1016/s1836-9553(10)70038-2. PMID 20482475
- [Background] Onishi T, Shimada K, Sunayama S, Ohmura H, Sumide T, Masaki Y, Fukao K, Nishitani M, Kume A, Sato H, Naito H, Kawai S, Amano A, Daida H. Effects of cardiac rehabilitation in patients with metabolic syndrome after coronary artery bypass grafting. J Cardiol. 2009 Jun;53(3):381-7. doi: 10.1016/j.jjcc.2009.01.004. Epub 2009 Feb 23. PMID 19477380
- [Background] Sumide T, Shimada K, Ohmura H, Onishi T, Kawakami K, Masaki Y, Fukao K, Nishitani M, Kume A, Sato H, Sunayama S, Kawai S, Shimada A, Yamamoto T, Kikuchi K, Amano A, Daida H. Relationship between exercise tolerance and muscle strength following cardiac rehabilitation: comparison of patients after cardiac surgery and patients with myocardial infarction. J Cardiol. 2009 Oct;54(2):273-81. doi: 10.1016/j.jjcc.2009.05.016. PMID 19782265
- [Background] Adams J, Lotshaw A, Exum E, Campbell M, Spranger CB, Beveridge J, Baker S, McCray S, Bilbrey T, Shock T, Lawrence A, Hamman BL, Schussler JM. An alternative approach to prescribing sternal precautions after median sternotomy, "Keep Your Move in the Tube". Proc (Bayl Univ Med Cent). 2016 Jan;29(1):97-100. doi: 10.1080/08998280.2016.11929379. PMID 26722187
- [Background] El-Ansary D, LaPier TK, Adams J, Gach R, Triano S, Katijjahbe MA, Hirschhorn AD, Mungovan SF, Lotshaw A, Cahalin LP. An Evidence-Based Perspective on Movement and Activity Following Median Sternotomy. Phys Ther. 2019 Dec 16;99(12):1587-1601. doi: 10.1093/ptj/pzz126. PMID 31504913
- [Background] Katijjahbe MA, Granger CL, Denehy L, Royse A, Royse C, Bates R, Logie S, Nur Ayub MA, Clarke S, El-Ansary D. Standard restrictive sternal precautions and modified sternal precautions had similar effects in people after cardiac surgery via median sternotomy ('SMART' Trial): a randomised trial. J Physiother. 2018 Apr;64(2):97-106. doi: 10.1016/j.jphys.2018.02.013. Epub 2018 Mar 27. PMID 29602750
- [Background] Mungovan SF, Singh P, Gass GC, Smart NA, Hirschhorn AD. Effect of physical activity in the first five days after cardiac surgery. J Rehabil Med. 2017 Jan 19;49(1):71-77. doi: 10.2340/16501977-2165. PMID 28101566
- [Background] Ennis S, Lobley G, Worrall S, Evans B, Kimani PK, Khan A, Powell R, Banerjee P, Barker T, McGregor G. Effectiveness and Safety of Early Initiation of Poststernotomy Cardiac Rehabilitation Exercise Training: The SCAR Randomized Clinical Trial. JAMA Cardiol. 2022 Aug 1;7(8):817-824. doi: 10.1001/jamacardio.2022.1651. PMID 35731506